CLINICAL TRIAL: NCT02756403
Title: A Randomized Controlled Trial of Three Prophylactic Antibiotic Regimens for First Trimester Surgical Abortion
Brief Title: A Randomized Controlled Trial of Three Antibiotic Regimens for First Trimester Abortions
Status: Completed | Phase: Not Applicable | Type: Interventional
Sponsor: Medstar Health Research Institute (Other)
Collaborators: Society of Family Planning (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Single Group | Masking: Triple | Purpose: Prevention
Other Study IDs: 2015-159
Record Dates: First submitted 2016-03-20; First posted 2016-04-29 (Estimated); Results first posted 2022-02-11 (Actual); Last update posted 2022-02-11 (Actual); Status verified 2022-02

CONDITIONS: First Trimester Abortion
MeSH Terms: interventions — Azithromycin; Doxycycline; Metronidazole

STUDY DESIGN:
Who Masked: Participant, Care Provider, Investigator
Oversight: Data Monitoring Committee: No

ARMS (4):
- Azithromycin (Active Comparator): 500 mg of Azithromycin
  Interventions: Drug: Azithromycin
- Doxycycline (Active Comparator): 200 mg of Doxycycline
  Interventions: Drug: Doxycycline
- Metronidazole (Active Comparator): 500 mg of Metronidazole
  Interventions: Drug: Metronidazole
- Placebo (Placebo Comparator): Inactive Ingredient
  Interventions: Drug: Placebo

INTERVENTIONS:
Drug: Azithromycin — 500 mg
  Arms: Azithromycin
Drug: Doxycycline — 200 mg
  Arms: Doxycycline
Drug: Metronidazole — 500 mg
  Arms: Metronidazole
Drug: Placebo — Placebo pills will be given before the uterine aspiration. Antibiotics will be given after the uterine aspiration.
  Arms: Placebo

SUMMARY:
This study, a double blinded randomized controlled trial, is being done to compare side effects of commonly used antibiotic regimens prior to same day abortion procedures.

In total, 180 pregnant women in their first trimester of pregnancy (5 0/6-13 6/7 weeks gestation) will be randomized to receive one of the three commonly used antibiotics (azithromycin, doxycycline, metronidazole) for same day abortion procedures or placebo prior to their abortion procedure. Approximately, 30-60 mins after study drug administration, the procedure will be performed.

A sub-study will be completed on 40 women who consent to endometrial sampling and to have their blood drawn.

DETAILED DESCRIPTION:
Main Study:

Women will be randomized to receive single oral doses of azithromycin 500 mg, doxycycline 200 mg, metronidazole 500 mg, or placebo. Computer-generated randomization will be used to assign participants to one of the four treatment arms. Women receiving placebo will receive antibiotic prophylaxis after completion of the study.

Both the participants and the investigators will be blinded as to the treatment group. This will be accomplished by placing the study medication inside opaque gelatin capsules. We will randomize participants by assigning them to the next of the sequentially numbered sealed opaque study packets, containing the gelatin capsules with study medication inside. A second envelope will be opened after completion of all study procedure and will only say if the participant received placebo, so that additional antibiotics can be given.

Participants will swallow the appropriate medication approximately 30-60 minutes prior to the surgical abortion (15-90 minutes range is acceptable). Study population will be all eligible patients undergoing surgical abortion in the first trimester at Washington Hospital Center and Planned Parenthood Metropolitan Washington. We will assess pain and side effects via written questionnaire at three different time points throughout the day, once at time of consent, before and after the procedure. Patients will be contacted within 1-2 weeks for follow-up and again pain and side effects will be assessed, as well.

Sub-study:

Forty (n=40) women will be recruited to undergo immediate post-procedure endometrial sampling. Sub-study patients will have a blood sample collected via venipuncture before leaving the procedure room, as well. No testing will be performed for participants receiving placebo.

The primary objective is to determine if the side effects associated with individual medications are more similar to placebo than the others.

The sub-study aims to explore our ability to identify bacteria within the uterine cavity. The objective is to assess the feasibility of identifying bacteria within the uterus after abortion.

ELIGIBILITY:
Inclusion Criteria:

* Women in good general health.
* English speaking.
* Age 18 or over.
* Seeking non-urgent surgical termination of pregnancy.
* Gestational age of 5 0/7 to 13 6/7 weeks, confirmed by sonogram.

Exclusion Criteria:

* Less than 18 years of age.
* Early pregnancy failure or fetal demise.
* Poor general health that would prevent one from tolerating the medication or surgical procedure.
* Intolerance, allergy, or contraindication to any of the study medications.
* Inability to tolerate oral intake due to current nausea or vomiting.
* Diagnosis of hyperemesis gravidarum with current pregnancy.
* Need of an urgent surgical abortion.
* Gestational age outside of 5-13 6/7 weeks by sonogram.

Min Age: 18 Years | Sex: Female | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 181 (Actual)
Dates: Start 2016-03; Primary Completion 2017-07 (Actual); Study Completion 2017-07 (Actual)

CONTACTS AND LOCATIONS:
Locations (2):
- United States (2):
  - MedStar Washington Hospital Center, Washington D.C., District of Columbia
  - Planned Parenthood Metropolitan Washington, Silver Spring, Maryland

IPD SHARING:
Plan to Share IPD: No

RESULTS

PARTICIPANT FLOW:
Period: Overall Study
Arm/Group | Azithromycin | Doxycycline | Metronidazole | Placebo
Started | 46 | 45 | 43 | 47
Completed | 46 | 42 | 41 | 45
Not Completed | 0 | 3 | 2 | 2
Not completed — Unable to swallow medication | 0 | 1 | 1 | 1
Not completed — Did not complete Procedure | 0 | 1 | 0 | 0
Not completed — Changed Mind About Procedure | 0 | 0 | 1 | 0
Not completed — Protocol Violation | 0 | 1 | 0 | 1

BASELINE CHARACTERISTICS:
Population: 2 Patients excluded for protocol violations, 2 withdrawn due to cancelled Abortion procedures, 3 withdrawn as unable to tolerate study medications.
Groups:
- Total: Total of all reporting groups
Arm/Group | Azithromycin | Doxycycline | Metronidazole | Placebo | Total
Number analyzed (Participants) | 46 | 42 | 41 | 45 | 174
Age, Continuous [Mean (Standard Deviation); unit: years] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  years | 25.1 (5.0) | 26.2 (6.4) | 26.5 (5.5) | 28.6 (6.1) | 26.6 (5.9)
Sex: Female, Male [Count of Participants; unit: Participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  Participants
    Female | 46 | 42 | 41 | 45 | 174
    Male | 0 | 0 | 0 | 0 | 0
Race (NIH/OMB) [Count of Participants; unit: Participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  Participants
    American Indian or Alaska Native | 0 | 0 | 0 | 0 | 0
    Asian | 2 | 0 | 1 | 2 | 5
    Native Hawaiian or Other Pacific Islander | 0 | 0 | 0 | 0 | 0
    Black or African American | 29 | 31 | 27 | 34 | 121
    White | 7 | 6 | 7 | 4 | 24
    More than one race | 7 | 4 | 4 | 5 | 20
    Unknown or Not Reported | 1 | 1 | 2 | 0 | 4
BMI [Mean (Standard Deviation); unit: kg/m^2] — Body Mass Index Population: Excluded protocol violations and patients unable to complete study, see Patient Flow. Unable to measure height/weight for one immobilized patient (metronidazole group)
  kg/m^2 | 27.8 (6.2) | 27.0 (7.3) | 29.5 (8.5) | 29.0 (7.0) | 28.3 (7.3)
Education [Count of Participants; unit: Participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  Participants
    Less than High School | 4 | 0 | 3 | 0 | 7
    HS Grad or Equivalent | 17 | 16 | 13 | 16 | 62
    Some College | 14 | 18 | 20 | 17 | 69
    College Grad | 9 | 5 | 4 | 10 | 28
    Graduate School | 2 | 3 | 1 | 2 | 8
Parous [Count of Participants; unit: Participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  Participants
    Nulliparous | 21 | 17 | 10 | 17 | 65
    Parous | 25 | 25 | 31 | 28 | 109
Marital Status [Count of Participants; unit: Participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  Participants
    Single | 36 | 31 | 34 | 31 | 132
    Married | 4 | 9 | 3 | 5 | 21
    Divorced | 0 | 1 | 1 | 3 | 5
    Separated | 0 | 0 | 0 | 2 | 2
    Cohabitating | 6 | 1 | 3 | 4 | 14
Work Status [Number; unit: participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow.
  Several patients indicated multiple answers
  participants
    Full Time Work: number analyzed (Participants) | 46 | 41 | 40 | 45 | 172
    Full Time Work | 20 | 19 | 16 | 23 | 78
    Part Time Work | 8 | 6 | 9 | 10 | 33
    Full Time Student | 4 | 5 | 4 | 4 | 17
    Unemployed | 14 | 13 | 11 | 6 | 44
    Homemaker | 0 | 1 | 1 | 1 | 3
    Other | 0 | 0 | 0 | 1 | 1
Prior Abortion [Count of Participants; unit: Participants] — Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  Participants
    Yes | 21 | 21 | 26 | 34 | 102
    No | 25 | 21 | 15 | 11 | 72
Gestational age [Mean (Standard Deviation); unit: days] — at time of procedure, by ultrasound criteria Population: Excluded protocol violations and patients unable to complete study, see Patient Flow
  days | 60.9 (16.8) | 63.9 (17.1) | 65 (12.2) | 67.5 (15.8) | 64.3 (15.7)

OUTCOME MEASURES:

1. Primary Outcome: Nausea Scale
Description: Nausea symptom was collected at different time points via surveys (None, Mild, Moderate, Severe)
Time Frame: 1 Day
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Doxycycline | Metronidazole | Placebo
Number analyzed (Participants) | 46 | 42 | 41 | 45
Participants
  Baseline: None | 8 | 9 | 6 | 6
  Baseline: Mild | 18 | 15 | 10 | 14
  Baseline: Moderate | 13 | 11 | 20 | 16
  Baseline: Severe | 7 | 7 | 5 | 9
  Before Procedure: None | 34 | 36 | 36 | 39
  Before Procedure: Mild | 8 | 4 | 5 | 5
  Before Procedure: Moderate | 2 | 2 | 0 | 0
  Before Procedure: Severe | 2 | 0 | 0 | 1
  After Procedure: None | 35 | 28 | 34 | 37
  After Procedure: Mild | 7 | 5 | 6 | 8
  After Procedure: Moderate | 4 | 6 | 1 | 0
  After Procedure: Severe | 0 | 3 | 0 | 0

2. Primary Outcome: Emesis Severity
Description: Emesis severity assessment collected at different time points (None, Mild, Moderate, Severe)
Time Frame: 1 Day
Population: 4 Subjects failed to complete the entire post-procedure survey: 1 Azithromycin group, 2 in Metronidazole group, 1 in Placebo group
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Doxycycline | Metronidazole | Placebo
Number analyzed (Participants) | 46 | 42 | 41 | 45
Participants
  Baseline: None | 20 | 24 | 13 | 17
  Baseline: Mild | 12 | 8 | 16 | 15
  Baseline: Moderate | 6 | 6 | 11 | 8
  Baseline: Severe | 8 | 4 | 1 | 5
  Before Procedure: None | 43 | 42 | 41 | 44
  Before Procedure: Mild | 1 | 0 | 0 | 1
  Before Procedure: Moderate | 2 | 0 | 0 | 0
  Before Procedure: Severe | 0 | 0 | 0 | 0
  After Procedure: number analyzed (Participants) | 45 | 42 | 39 | 44
  After Procedure: None | 42 | 35 | 39 | 44
  After Procedure: Mild | 2 | 1 | 0 | 0
  After Procedure: Moderate | 1 | 5 | 0 | 0
  After Procedure: Severe | 0 | 1 | 0 | 0

3. Secondary Outcome: Pain Scale
Description: Pain symptoms will be collected at different time points via surveys (None, Mild, Moderate, Severe)
Time Frame: Day 1
Population: 4 patients had incomplete post-procedure surveys: 1 in Azithromycin group, 2 in Metronidazole group, 1 in Placebo group
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Doxycycline | Metronidazole | Placebo
Number analyzed (Participants) | 46 | 42 | 41 | 45
Participants
  Baseline Pain: None | 20 | 17 | 16 | 13
  Baseline Pain: Mild | 18 | 14 | 16 | 18
  Baseline Pain: Moderate | 6 | 8 | 6 | 11
  Baseline Pain: Severe | 2 | 3 | 3 | 3
  Before Procedure: None | 35 | 38 | 35 | 39
  Before Procedure: Mild | 9 | 4 | 6 | 5
  Before Procedure: Moderate | 1 | 0 | 0 | 1
  Before Procedure: Severe | 1 | 0 | 0 | 0
  After Procedure: number analyzed (Participants) | 45 | 42 | 39 | 44
  After Procedure: None | 18 | 16 | 9 | 15
  After Procedure: Mild | 18 | 17 | 17 | 16
  After Procedure: Moderate | 6 | 7 | 12 | 11
  After Procedure: Severe | 3 | 2 | 1 | 2

4. Secondary Outcome: Serum Antibiotic Levels
Description: Serum antibiotic levels drawn at time of endometrial sampling in subset of patients
Time Frame: 3 hours
Population: Subset of patients who had serum antibiotic levels drawn
Measure: Mean (Standard Deviation); unit: mcg/mL
Arm/Group | Azithromycin | Doxycycline | Metronidazole
Number analyzed (Participants) | 5 | 6 | 8
mcg/mL | 0.41 (0.22) | 1.1 (0.8) | 8.2 (3.8)

5. Secondary Outcome: Endometrial Growth
Description: Endometrial Growth on non-selective, Staph Selective, Strep Selective, and Gram negative selective Agar
Time Frame: 3 Days
Population: Subset of patients with endometrial swab cultured
Measure: Count of Participants; unit: Participants
Arm/Group | Azithromycin | Doxycycline | Metronidazole | Placebo
Number analyzed (Participants) | 7 | 11 | 11 | 4
Participants
  No Growth | 4 | 7 | 8 | 1
  Trypic Soy Non-Selective Agar | 3 | 4 | 3 | 2
  Mannitol Salt Agar (Staph selective) | 1 | 2 | 0 | 1
  Streptococcus Agar (Strep selective) | 1 | 1 | 1 | 3
  MacConkey Agar (gram neg selective) | 0 | 0 | 0 | 0

ADVERSE EVENTS:
Time Frame: One week
Description: Patients involved in study were called on telephone at one week to assess for any adverse events.
Groups:
- Metronidazole: Patients receivingMetronidazole for preprocedure antibiotic
- Azithromycin: Patients receiving Azithromycin for preprocedure antibiotic
- Doxycycline: Patients receiving Doxycycline for preprocedure antibiotic
- Placebo: Patients receiving Placebo preprocedure
Arm/Group | Metronidazole | Azithromycin | Doxycycline | Placebo
All-Cause Mortality (participants affected / at risk) | 0/41 | 0/46 | 0/42 | 0/45
Serious Adverse Events (participants affected / at risk) | 1/41 | 0/46 | 0/42 | 0/45
Other Adverse Events (participants affected / at risk) | 0/41 | 0/46 | 0/42 | 0/45
SERIOUS ADVERSE EVENTS; cells are participants affected of the arm's N at risk (number of events):
Term (organ system) | Metronidazole (N=41) | Azithromycin (N=46) | Doxycycline (N=42) | Placebo (N=45)
Inpatient Hospitalization (Pregnancy, puerperium and perinatal conditions) | 1 (1) | 0 (0) | 0 (0) | 0 (0)

CERTAIN AGREEMENTS:
Principal investigators are sponsor employees: No; Agreement restricts PI disclosure of results: No

DOCUMENTS (1):
  • Study Protocol and Statistical Analysis Plan (2015-06-26): https://cdn.clinicaltrials.gov/large-docs/03/NCT02756403/Prot_SAP_000.pdf